CLINICAL TRIAL: NCT03839927
Title: Validity and Reliability of the Turkish Version of The Life-Space Assessment Scale
Brief Title: Turkish Version of The Life-Space Assessment Scale
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, PT.MSc, Firat University
Other Study IDs: FiratU
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Physical Activity
Keywords: Life Space Assesment; Daily Life Activity; Geriatrics; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation Group: Survey Application
  Interventions: Other: Validity and reliability of Life-Space Assesment

INTERVENTIONS:
Other: Validity and reliability of Life-Space Assesment — Life-Space Assesment and SF-36 surveys will be applied. The reliability and validity of the results will be analyzed.

SUMMARY:
In mobility, the potential for mobility and social inclusion, according to individual desires, represents the primary component of well-being and should be a priority for caregivers of older adults and older adults. As a result of our literature researches, it was found that there was no Turkish scale evaluating the living area. For this reason, this study was planned in order to translate the Turkish Life-Space Assessment [LSA] into Turkish, to investigate the validity and reliability of the Turkish version and to perform its cultural adaptation. Our study is expected to improve the quality of health assessment in our country, to contribute to objective evaluation methods, and to provide benefits such as assisting physicians, physiotherapists and other related health care team during the evaluation process.

DETAILED DESCRIPTION:
Decrease in movement and limitation is common in older adults. Compared to the general population where mobility is restricted in 10.1% of individuals, this rate rises to 15.4% for those aged 50-69 and increases to 36.2% after 70 years of age . Mobility has direct and direct consequences for maintaining the independence and autonomy of all older adults. Decreased mobility increases both quality of life and formal and informal care needs . For older adults, mobility can be the most important functional skill required to maintain social roles and quests, and the decrease in mobility is often in front of disability in daily living activities (GYA) (2). Mobility assessments range from biomechanical measurements to broader assessments of people's daily lives .

Ambulation problems are fundamentally conceptualized in relation to internal and upper-level movement (when a person leaves his / her home or takes a mile of distance üst etc.). This limitation of movement is common among older adults and increases with age. The emergence and progression of age-related chronic diseases is a reason why the elderly population continues to be at increased risk for mobility loss.

Traditional measures such as GYA (bath, dressing, transfer, toilet and food) and Instrumental Activities of Daily Life (GYAA - light and heavy housework, food preparation, shopping and money management) are special functions that are an integral part of mobility. On the other hand, the living space reflects integration and social inclusion in geographically defined areas and measures how much, how often, and how independently individuals act in their environment. This assessment provides a measure of mobility throughout the observed function among elderly adults living in the community, which may have different and multiple chronic diseases and different disability levels. Living space mobility enables the participation of individuals in the community or the mobility of the individual.

While the maintenance of all aspects of health in aging individuals has gained importance as the focus of the research, there has been much debate about proper measurement. Muldoon et al. Reported that it is very important in the post-illness effects beyond the immediate effects of the disease to examine the effects of people on their daily lives. Traditional treatment and evaluation methods are focused on function and ability to perform certain tasks . However, the difficulty in these measures may not be evident until later in disability models. In contrast, the habitat provides a measure of full mobility continuity, which allows for differentiation in the upper limits of in healthy aging.

* The methodological model of the study is validity reliability study.
* The validity and reliability of Turkish LSA , whose validity and reliability have been demonstrated in different languages (French, English), will be investigated. Authorization from the author of the original LSA (Prof. Patricia SAWYER) was obtained.
* Hypotheses:

H1 1: The Turkish version of LSA is a valid scale. H1 2: The Turkish version of LSA is a reliable scale.

* It is planned that the data will be collected on a voluntary basis from the individuals who live in the province of Elazığ and comply with the inclusion criteria.
* In the validity and reliability studies, it is stated that the sample size should be at least five times or even ten times the number of items. Since LSA is a 20-item scale and the sample size is recommended as x5-x10 in similar studies, it is planned to carry out the study on 100 volunteer individuals .
* Inclusion Criteria of the Volunteers

  * 65 years and over,
  * Contactable,
  * Individuals who are independent in their daily activities.
* Criteria for Exclusion of Participants in Research

  * 64 years and under,
  * Do not read, understand and write in Turkish,
  * Unable to communicate,
  * Individuals dependent on one in daily living activities.

Age, gender, height, body weight, body mass index, marital status, working status, residence area (urban - rural), accessibility of the housing (fully accessible, partially accessible and not accessible) information about the life expectancy in the neighborhood, the history of falling within the last 6 months, the use of ancillary equipment, the existence of the driver's license, the existence of a single life, the education and income levels, and the information contained in the demographic information form.

In order to evaluate the quality of life of the participants in the study, the validity and reliability study developed by Ware in 1987 and in our country was reviewed by Koçyiğit et al. SF-36 scale was used. In this scale, where health is examined in 8 components, high scores indicate a better level of health. SF-36 scale; physical function (FF) (limitation in physical activity due to health problems), physical role (FR) (restriction in daily living activities due to health problems), bodily pain (BA), general health (GS) (assessment of health of the person in general), vitality ( CA) consists of general mental health (GRS), social functionality (SF), and emotional role (DR) (restriction of daily living activities due to mental health problems). The SF-36 scale scales 100 points and the scores vary between 0 and 100 points for each component .

The translation process for the preparation of the Turkish LSA form to be applied to the cases will include:

In order to translate the LSA into Turkish and to investigate its validity and reliability, the recommendations developed by Guillemin et al. And Beaton et al. Will be utilized . The English version of LSA will be translated into Turkish by two persons independently. These two different Turkish versions will be analyzed by an expert committee. The translations will be evaluated by considering Turkish cultural characteristics. A common version (Version1) will then be created from these translations. Version 1 will be translated back to English by a non-medical specialist and a native speaker. This will be compared with the original LSA by the expert committee to determine the equivalence of the reverse translation. At the end of this phase, the common version 2 will be obtained and compared with the original LSA to determine equivalence. A pilot study will be carried out with 20 participants (10 males and 10 females) after confirming the equivalence of the original LSA and Turkish version of the committee or, if necessary, making some corrections. The main objective of this phase is to determine whether participants understand the questions. The clarity and clarity of each item will be scored by the participants with the Likert scale and the Content Validity Index (CVI) of the LSA will be calculated. The Turkish version of the LSA will be reviewed by the expert committee in the light of the findings and minor changes will be made if necessary. Once the final decision has been made, the Turkish version of the LSA will be applied to the study population. To investigate the reliability of the scale, the test-retest procedure will be followed and the scale will be applied to the same participants for the second time in 24-hour intervals.

SPSS for Windows 20.00 computer package program will be used for all statistical analysis. Descriptive statistical information shall be given as mean ± standard deviation (x ± SD) or%. Interclass Correlation Coefficients (ICC) and Cronbach güvens coeffi for reliability and internal consistency of LSA

ELIGIBILITY:
Inclusion Criteria:

* 65 years and over,
* Contactable,
* Individuals who are independent in their daily activities

Exclusion Criteria:

* 64 years and under,
* Do not read, understand and write in Turkish,
* Unable to communicate,
* Individuals dependent on one in daily living activities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Turkey sample
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Life-Space Assesment | 3 Months
  Life Space Assessment is a scale that measures 5 different environments (such as in-house, neighborhood, out-of-province) and evaluates the amount and quality of movement in these environments.

SECONDARY OUTCOMES:
Short Form-36 | 3 Months
  In this scale, where health is examined in 8 components, high scores indicate a better level of health. SF-36 scale; physical functionality (restriction in physical activity due to health problems), physical role (restriction in activities of daily living due to health problems), physical pain, general health (assessment of health of the person in general), vitality, general mental health, social functionality and emotional role. The SF-36 scales are rated over 100 points and the scores vary between 0 and 100 points for each component.

IPD SHARING:
Plan to Share IPD: Undecided
Survey data Participant data

REFERENCES:
- [Background] Iezzoni LI, McCarthy EP, Davis RB, Siebens H. Mobility difficulties are not only a problem of old age. J Gen Intern Med. 2001 Apr;16(4):235-43. doi: 10.1046/j.1525-1497.2001.016004235.x. PMID 11318924
- [Background] Cesari M, Marzetti E, Canevelli M, Guaraldi G. Geriatric syndromes: How to treat. Virulence. 2017 Jul 4;8(5):577-585. doi: 10.1080/21505594.2016.1219445. Epub 2016 Aug 11. PMID 27540686
- [Background] Stewart CM, Wheeler TL 2nd, Markland AD, Straughn JM Jr, Richter HE. Life-space assessment in urogynecology and gynecological oncology surgery patients: a measure of perioperative mobility and function. J Am Geriatr Soc. 2009 Dec;57(12):2263-8. doi: 10.1111/j.1532-5415.2009.02557.x. Epub 2009 Oct 26. PMID 19874406
- [Background] Muldoon MF, Barger SD, Flory JD, Manuck SB. What are quality of life measurements measuring? BMJ. 1998 Feb 14;316(7130):542-5. doi: 10.1136/bmj.316.7130.542. No abstract available. PMID 9501721
- [Background] Peel C, Sawyer Baker P, Roth DL, Brown CJ, Brodner EV, Allman RM. Assessing mobility in older adults: the UAB Study of Aging Life-Space Assessment. Phys Ther. 2005 Oct;85(10):1008-119. PMID 16180950
- [Background] Hou WH, Yeh TS, Liang HW. Reliability and validity of the Taiwan Chinese version of the Lower Extremity Functional Scale. J Formos Med Assoc. 2014 May;113(5):313-20. doi: 10.1016/j.jfma.2012.07.032. Epub 2012 Sep 15. PMID 24746117
- [Background] Wright JG, Young NL. A comparison of different indices of responsiveness. J Clin Epidemiol. 1997 Mar;50(3):239-46. doi: 10.1016/s0895-4356(96)00373-3. PMID 9120522
- [Background] Auger C, Demers L, Gelinas I, Routhier F, Jutai J, Guerette C, Deruyter F. Development of a French-Canadian version of the Life-Space Assessment (LSA-F): content validity, reliability and applicability for power mobility device users. Disabil Rehabil Assist Technol. 2009 Jan;4(1):31-41. doi: 10.1080/17483100802543064. PMID 19172479
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Ayvat E, Kilinc M, Kirdi N. The Turkish version of the Physical Activity Scale for the Elderly (PASE): its cultural adaptation, validation, and reliability. Turk J Med Sci. 2017 Jun 12;47(3):908-915. doi: 10.3906/sag-1605-7. PMID 28618742
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Cacchio A, De Blasis E, Necozione S, Rosa F, Riddle DL, di Orio F, De Blasis D, Santilli V. The Italian version of the lower extremity functional scale was reliable, valid, and responsive. J Clin Epidemiol. 2010 May;63(5):550-7. doi: 10.1016/j.jclinepi.2009.08.001. Epub 2009 Nov 12. PMID 19913388
- [Background] Yeung TS, Wessel J, Stratford P, Macdermid J. Reliability, validity, and responsiveness of the lower extremity functional scale for inpatients of an orthopaedic rehabilitation ward. J Orthop Sports Phys Ther. 2009 Jun;39(6):468-77. doi: 10.2519/jospt.2009.2971. PMID 19487822